CLINICAL TRIAL: NCT06165276
Title: Phase I Study of the Safety and Immunogenicity of a Quadrivalent Meningococcal (A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine in Adults, Toddlers, and Infants
Brief Title: A Phase I, Randomized, Modified Single-blind, Active-controlled (Infants Only), Four-stage, Step-down, Comparative, Multi-center Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MET28
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: Meningococcal Immunization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1 (Experimental): Adults receiving Low Dose TetraMen-T with adjuvant
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine (TetraMen-T).
- Group 2 (Experimental): Adults receiving High Dose TetraMen-T without adjuvant
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine (TetraMen-T).
- Group 3 (Experimental): Toddlers receiving Low Dose TetraMen-T with adjuvant
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine (TetraMen-T).
- Group 4 (Experimental): Toddlers receiving High Dose TetraMen-T without adjuvant
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine (TetraMen-T).
- Group 5 (Experimental): Infants receiving Low Dose TetraMen-T with adjuvant. Subjects were to receive a booster dose of the same formulation at age 13 months
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine (TetraMen-T).
- Group 6 (Experimental): Infants receiving Low Dose TetraMen-T with adjuvant. Subjects were to receive a booster dose of the same formulation at age 13 months
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine (TetraMen-T).
- Group 7 (Experimental): Infants receiving High Dose TetraMen-T without adjuvant. Subjects were to receive a booster dose of the same formulation at age 13 months
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine (TetraMen-T).
- Group 8 (Active Comparator): Infants receiving Menjugate ®. Subjects were to receive a booster dose of low-dose adjuvanted TetraMen-T at age 13 months. Routine vaccines were deferred.
  Interventions: Biological: Meningococcal Group C-CRM197 Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Tetanus Protein Conjugate Vaccine (TetraMen-T). — Pharmaceutical form:suspension for injection-Route of administration:Intramuscular (IM)
  Other Names: 395
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7
Biological: Meningococcal Group C-CRM197 Conjugate Vaccine — Pharmaceutical form:suspension for injection-Route of administration:Intramuscular (IM)
  Other Names: Menjugate®
  Arms: Group 8

SUMMARY:
The study will include groups of adults, toddlers, and infants who will receive different formulations of TetraMen-T, and one group of infants who will receive a control vaccine, Menjugate®. The primary objectives and their endpoints will be assessed in infants who receive TetraMen-T. The secondary objectives and their endpoints will be assessed only in the subset of infants who receive a booster dose of TetraMen-T.

Primary objectives:

1. To describe the safety profile in infants following three injections of TetraMen-T, either a low-dose formulation (2 µg olysaccharide per serogroup without adjuvant), a low-dose adjuvanted formulation (2 µg polysaccharide per serogroup with djuvant), or a high-dose formulation (10 µg polysaccharide per serogroup without adjuvant), administered concomitantly with routine vaccines (Pentacel®, Prevnar®, and Engerix-B®).
2. To describe the immunogenicity profile in infants following three injections of TetraMen-T, either a low-dose formulation (2 µg polysaccharide per serogroup without adjuvant), a low-dose adjuvanted formulation (2 µg polysaccharide per serogroup with adjuvant), or a high-dose formulation (10 µg polysaccharide per serogroup without adjuvant), administered on comitantly with routine vaccines (Pentacel®, Prevnar®, and Engerix-B®).

Secondary objectives:

1. To describe the safety profile in a subset of infants following a booster dose of TetraMen-T, either a low-dose formulation (2 µg polysaccharide per serogroup without adjuvant), a low-dose adjuvanted formulation (2 µg polysaccharide per erogroup with adjuvant), or a high-dose formulation (10 µg polysaccharide per serogroup without adjuvant), at 13 months of age.
2. To describe the immunogenicity profile in a subset of infants following a booster dose of TetraMen-T, either a low-dose formulation (2 µg polysaccharide per serogroup without adjuvant), a low-dose adjuvanted formulation (2 µg polysaccharide per serogroup with adjuvant), or a high-dose formulation (10 µg polysaccharide per serogroup without adjuvant), at 13 months of age.

DETAILED DESCRIPTION:
Up to 24 months

ELIGIBILITY:
Inclusion Criteria: -Subject is healthy, as determined by medical history and physical assessment.

-At the time of vaccination on Day 0, subject was the following age: Adults: aged ≥18 to < 40 years Toddlers: aged ≥12 to < 19 months Infants: aged 2 months + 28 days (60 to 88 days)

* Institutional Review Board (IRB)-approved informed consent form signed by the subject or the subject's parent/legal guardian. Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 60 Days to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 285 (Actual)
Dates: Start 2006-07-25 (Actual); Primary Completion 2008-08-27 (Actual); Study Completion 2008-08-27 (Actual)

PRIMARY OUTCOMES:
Presence of solicited injection site reactions (ie, prelisted in the participant's diary card [DC] and in the electronic case report form [eCRF]) occurring up to 7 days after injection | Up to 7 days after injection
Presence of any unsolicited systemic adverse events (AEs) reported up to 28 days after injection | Up to 28 days after injection
Presence of serious adverse events (SAEs) throughout the trial. | From baseline up to 24 months
Incidence of treatment-emergent antibodies responses | From baseline up to 24 months

SECONDARY OUTCOMES:
After booster dose of TetraMen-T: Presence of solicited injection site reactions (ie, prelisted in the participant's diary card [DC] and in the electronic case report form [eCRF]) occurring up to 7 days after injection | Up to 7 days after injection
After booster dose of TetraMen-T: Presence of any unsolicited systemic adverse events (AEs) reported up to 28 days after injection | Up to 28 days after injection
After booster dose of TetraMen-T: Presence of serious adverse events (SAEs) throughout the trial. | From baseline up to 24 months
After booster dose of TetraMen-T: Incidence of treatment-emergent antibodies responses | From baseline up to 24 months